CLINICAL TRIAL: NCT07007052
Title: Open Label Phase II Study Evaluating the Efficacy and Safety of the Combination of Tagraxofusp and Venetoclax in Treatment-naive Blastic Plasmacytoid Dendritic Cell Neoplasm Patients
Brief Title: Phase II Study Evaluating the Efficacy and Safety of the Combination of Tagraxofusp and Venetoclax in Treatment-naive Blastic Plasmacytoid Dendritic Cell Neoplasm Patients
Acronym: TAGVEN
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: French Innovative Leukemia Organisation (Other)
Collaborators: Stemline Therapeutics, Inc. (Industry); AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAGVEN
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Blastic Plasmacytoid Dendritic Cell Neoplasm (BPDCN)
Keywords: blastic plasmacytoid dendritic cell neoplasm; Combination of venetoclax + tagraxofusp; Composite complete remission; Complete remission; Evaluation of response
MeSH Terms: conditions — Blastic Plasmacytoid Dendritic Cell Neoplasm; Pathologic Complete Response | interventions — venetoclax; tagraxofusp

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single interventional arm (Experimental): For each 28 days-cycle of treatment :
  * venetoclax 400mg/day orally after a ramp-up period of 3-days
  * tagraxofusp starting at the end of the venetoclax ramp-up period i.e. at day 4 for twelve 28-days cycles, 12 μg/kg body weight administered as an intravenous infusion over 15 minutes, once daily, on days 1-3 of each cycle
  Interventions: Drug: Venetoclax; Drug: Tagraxofusp

INTERVENTIONS:
Drug: Venetoclax — Single interventional arm
  Other Names: ABT-199; GDC-0199; RG7601; selective BCL-2 inhibitor
Drug: Tagraxofusp — Single interventional arm
  Other Names: SL-401; CD123-directed cytotoxin

SUMMARY:
The goal of this clinical trial is to study the efficacy of the tagraxofusp + venetoclax combination in treatment-naive blastic plasmacytoid dendritic cell neoplasm adult patients.

The main question is to verify the response in patients after 3 cycles of tagraxofusp+venetolax and to demonstrate if the combination of tagraxofusp + venetoclax increases the rate of complete remission, assessed after 3 months of treatment.

Patients will receive a ramp-up phase of venetoclax during 3 days and at least 3 cycles of venetoclax. After, the investigators will evaluate the response, and depending on the response observed, patients may receive additional cycles of treatment for a maximum of 24 cycles, or receive an allograft or discontinue the treatment in the case of therapeutic failure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a confirmed BPDCN diagnosis according to WHO 2022 revised criteria and have not received previous treatment : patients with skin or lymph node lesions but no bone marrow involvement can be included
2. Age >18 years
3. Ability to understand the protocol and to sign an informed consent
4. Possibility of follow-up
5. ECOG < 3
6. Adequate renal function as demonstrated by a calculated creatinine clearance ≥ 60 mL/min by the Cockcroft-Gault formula.
7. Adequate cardiac function defined by LVEF >/= 50% by MUGA or ECHO and no clinically significant abnormalities on a 12-lead ECG
8. Albumin level≥3,2g/dL
9. Adequate liver function as demonstrated by:

   * aspartate aminotransferase (AST) ≤ 2.5 × ULN*
   * alanine aminotransferase (ALT) ≤ 2.5 × ULN*
   * bilirubin ≤ 3.0 × ULN, unless due to Gilbert's syndrome* * Unless considered due to leukemic organ involvement, in that cases values must be ≤ 10 × ULN
10. Men, and women of childbearing potential must be using a highly effective method of contraception
11. Negative urine/blood pregnancy test within 1 week prior to the initiation of treatment (if applicable)
12. Patient covered by any social security system

Exclusion Criteria:

1. Participation to another clinical trial with any investigative drug within 30 days prior to study enrolment.
2. Previous treatment with venetoclax or tagraxofusp
3. Treatment of BPDCN with any prior chemotherapy or investigational agents, except hydroxyurea for less than 14 days at the time of inclusion
4. Concomitant immunosuppressive therapy -except for low-dose prednisone (≤10 mg/day)
5. Known allergy or sensitivity to tagraxofusp, venetoclax, and any of its components or excipients.
6. Pregnant or breastfeeding woman
7. Known positivity for hepatitis B or C infection except for those subjects with an undetectable viral load or subjects with serologic evidence of prior vaccination to HBV
8. Evidence of uncontrolled systemic infection requiring therapy (viral, bacterial, or fungal)
9. Subject has any history of clinically significant condition(s) that in the opinion of the investigator would adversely affect his/her participating in this study including, but not limited to:

   * Cardiovascular disease e.g., NYHA heart failure > class 2, uncontrolled angina, history of myocardial infarction, unstable angina, or stroke within 6 months prior to study entry, uncontrolled hypertension, or clinically significant arrythmias not controlled by medication.
   * Renal, pulmonary, neurologic, psychiatric, endocrinologic, metabolic, immunologic, hepatic, cardiovascular disease, or bleeding disorder independent of leukemia.
10. Subject with a history of other malignancies within the last three years prior to study entry, except for:

    * Adequately treated in situ carcinoma of the breast or cervix uteri
    * Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin
    * Prostate cancer without needs for specific therapy
    * Previous malignancy confined and surgically resected (or treated with other modalities) with curative intent.
11. Malabsorption syndrome or other conditions that preclude enteral route of administration
12. Patient with hereditary fructose intolerance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2031-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who achieve a cCR (CR or Cri or CRc) after 3 TAGVEN cycles | From enrollment to the end of the third 28 days-cycle
  Evaluation will be done with a bone marrow aspirate, cytogenetics, metabolic imaging, study of MRD by NGS and flow-cytometry and SWAT SCORE

CONTACTS AND LOCATIONS:
Locations (34):
- France (34):
  - AMIENS - CH Amiens Picardie Site Sud, Amiens
  - ANGERS - CHU - Maladies du sang, Angers
  - ARGENTEUIL - Centre hospitalier Victor Dupouy, Argenteuil
  - AVIGNON - Centre Hospitalier, Avignon
  - BESANCON - Hôpital Jean Minjoz - Hématologie, Besançon
  - CLAMART - Hôpital d'Instruction des Armées de Percy, Clamart
  - Clermont-Ferrand - Chu Estaing, Clermont-Ferrand
  - Corbeil-Essonnes - Ch Sud Francilien, Corbeil-Essonnes
  - AP-HP- CRETEIL - CHU Henri Mondor, Créteil
  - Grenoble CHU - Hématologie Clinique, Grenoble
  - LILLE CHU - Hôpital Claude Huriez, Lille
  - Limoges CHU, Limoges
  - LYON HCL- Site Sud, Lyon
  - MARSEILLE - Institut Paoli-Calmettes, Marseille
  - METZ - CHR Metz-Thionville, Metz
  - Montpellier - Chu Saint Eloi, Montpellier
  - MULHOUSE GHRMSA - Hôpital E. Muller - Hématologie, Mulhouse
  - NANTES - Hôpital Hôtel Dieu - Hématologie Clinique, Nantes
  - Nimes CHU, Nîmes
  - APHP - Hôpital Saint-Louis - Hématologie adultes, Paris
  - APHP - HOPITAL COCHIN - Hématologie, Paris
  - AP-HP - Hôpital Necker, Paris
  - BORDEAUX - Hôpital Haut-Levêque, Pessac
  - POITIERS - Hôpital La Milétrie - Hématologie Clinique, Poitiers
  - REIMS - Hôpital Robert Debré - Hématologie Clinique, Reims
  - RENNES - CHU Pontchaillou - Hématologie Clinique, Rennes
  - ROUEN - Centre Henri Becquerel - Service Hématologie Clinique, Rouen
  - CHU SAINT-ETIENNE - iCHUSE, Saint-Etienne
  - Strasbourg - Institut de Cancerologie Strasbourg, Strasbourg
  - Toulouse - IUCT Oncopole - Service d'Hématologie, Toulouse
  - TOURS - Hôpital Bretonneau, Tours
  - NANCY - CHU de Brabois, Vandœuvre-lès-Nancy
  - VERSAILLES - Hôpital André Mignot, Versailles
  - Villejuif Igr - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No
The individual participant data collected will be analyzed by the sponsor and therefore not shared.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-15): https://cdn.clinicaltrials.gov/large-docs/52/NCT07007052/Prot_SAP_001.pdf